CLINICAL TRIAL: NCT05035095
Title: Efficacy and Safety of Oral Semaglutide 50 mg Once Daily in Subjects With Overweight or Obesity (OASIS 1)
Brief Title: Research Study to Investigate How Well Semaglutide Tablets Taken Once Daily Work in People Who Are Overweight or Living With Obesity (OASIS 1)
Acronym: OASIS 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9932-4737; U1111-1253-1670 (Other: World Health Organization (WHO)); 2020-002953-11 (EudraCT Number)
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral semaglutide (Experimental): Participants will receive once daily semaglutide tables in a dose escalating manner for 68 weeks: 3 mg (week 1-4), 7 mg (week 5-8), 14 mg (week 9-12), 25 mg (week 13-16) and 50 mg (week 17-68)
  Interventions: Drug: Oral semaglutide
- Oral semaglutide placebo (Placebo Comparator): All participants are given once daily dose for 68 weeks
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Oral semaglutide — Participants will receive a daily dose of oral semaglutide.
  Arms: Oral semaglutide
Drug: Placebo (semaglutide) — Oral placebo (semaglutide) once daily. Planned treatment duration will be 68 weeks.
  Arms: Oral semaglutide placebo

SUMMARY:
This study is being conducted to see if semaglutide tablets can be used as a treatment to help people living with overweight or obesity lose weight.

This study will look at the change in participants body weight. Participants will either get semaglutide tablets (new medicine) or placebo tablets ('dummy' medicine that looks like semaglutide but has no effect on the body). For a fair comparison, people are divided into two groups at random by a computer. This process is called randomisation.

Semaglutide tablets are new medicine being tested to treat overweight and obesity. Doctors in many countries can already prescribe semaglutide tablets at lower doses to treat type 2 diabetes.

Participants will get semaglutide or placebo tablets for 68 weeks and will need to take 1 tablet every morning

In addition to taking the medicine, participants will have talks with study staff about:

* healthy food choices
* how to be more physically active
* what participants can do to lose weight The study will last for about 1½ year.Participants will have 14 clinic visits and 7 phone calls with the study doctor. Blood samples will be taken at 10 visits.

Participants will have a test to check their heart done at 3 visits. Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period. If participant is a woman and is able to become pregnant, participant will be checked for pregnancy via urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Body mass index (BMI):

greater than or equal to 27.0 kg/m^2 with the presence of at least one of the following weight-related complications (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease OR greater than or equal to 30.0 kg/m^2

* History of at least one self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* HbA1c greater than or equal to 6.5% (48 mmol/mol) as measured by the central laboratory at screening
* A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  percentage-point
Achievement of body weight reduction greater than or equal to 5% (Yes/No) | At end-of-treatment (week 68)
  Count of participants

SECONDARY OUTCOMES:
Achievement of body weight reduction greater than or equal to 10% (Yes/No) | At end of treatment (week 68)
  Count of participants
Change in Short Form-36 (SF-36) Physical Function | From baseline (week 0) to end of treatment (week 68)
  Score points
Change in IWQOL-Lite-CT Physical Function | From baseline (week 0) to end of treatment (week 68)
  Score points
Change in waist circumference | From baseline (week 0) to end of treatment (week 68)
  measured in cm
Achievement of body weight reduction greater than or equal to 15% (Yes/No) | At end of treatment (week 68)
  Count of participants
Achievement of body weight reduction greater than or equal to 20% (Yes/No) | At end of treatment (week 68)
  Count of participants
Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 68)
  measured in kg/m^2
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 68)
  measured in mmHg
Change in diastolic blood pressure | From randomisation (week 0) to end of treatment (week 68)
  measured in mmHg
Change in HbA1c (glycated haemoglobin) | From baseline (week 0) to end of treatment (week 68)
  percentage-point
Change in fasting plasma glucose (FPG) | From baseline (week 0) to end of treatment (week 68)
  measured in mg/dL
Change in fasting serum insulin | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: Total cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: HDL (high density lipoprotein) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: LDL (low-density lipoprotein) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: VLDL (very-low density lipoprotein) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: Triglycerides | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in lipids: Free fatty acids | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Change in high sensitivity C-Reactive Protein | From baseline (week 0) to end of treatment (week 68)
  Ratio to baseline
Number of treatment emergent adverse events | From baseline (week 0) to end-of-trial (week 75)
  Count of events
Number of serious adverse events | From baseline (week 0) to end-of-trial (week 75)
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (56):
- United States (13):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - The Chappel Group Research, Kissimmee, Florida
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - East West Med Res Inst, Honolulu, Hawaii
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - Rochester Clinical Research, Inc., Rochester, New York
  - Accellacare, Wilmington, North Carolina
  - The University of Penn Center, Philadelphia, Pennsylvania
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Canada (5):
  - Ocean West Research Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
- Denmark (4):
  - Center for Klinisk Metabolisk Forskning, Hellerup
  - Hvidovre Hospital Endokrinologisk forsknings afsnit 159, Hvidovre
  - Sjællands Universitetshospital, Køge - Medicinsk Afdeling, Køge
  - Slagelse Sygehus Ambulatorium for hjertesygdomme, Slagelse
- Finland (3):
  - Obesity Research Unit, Helsinki
  - StudyCor, Jyväskylä
  - Seinäjoen keskussairaala, Seinäjoki
- France (7):
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Fondation Hôtel-Dieu, Le Creusot
  - Groupe Sos Sante-Hopital Le Creusot-Hotel Dieu-2, Le Creusot
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque-2, Pessac
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-2, Toulouse
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (8):
  - InnoDiab Forschung GmbH, Essen
  - Praxis Dr. med. M. Esser, Essen
  - Diabetes Zentrum Wandsbek Berufsausuebungsgemeinschaft GbR, Hamburg
  - Milek, Hohenmölsen, Hohenmölsen
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
  - MZM Praxis Drs. Erlinger, Stuttgart
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- Japan (3):
  - Chiba University Hospital_Diabetes, Metabolism and Endocrinology, Chiba-shi, Chiba
  - Suidoubashi Medical Clinic, Chiyoda-ku, Tokyo
  - Higashi-shinjuku clinic, Tokyo
- Poland (5):
  - NZOZ Przychodnia Specjalistyczna Medica, Lublin, Lubelski
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - Centrum Zdrowia Metabolicznego, Poznan, Wielkopolskie Voivodeship
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
- Russia (8):
  - Tumen State Medical University, Tyumen, Russia
  - LLC "Clinic of new technologies in Medicine", Dzerzhinskiy
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - Endocrinological Dispensary of Department of healthcare ser., Moscow
  - Federal Bureau for Medical and Social Expertise, Moscow
  - Joint Stock Company "Polyclinic Complex", Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Joint Stock Company "Medical technologies", Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Knop FK, Aroda VR, do Vale RD, Holst-Hansen T, Laursen PN, Rosenstock J, Rubino DM, Garvey WT; OASIS 1 Investigators. Oral semaglutide 50 mg taken once per day in adults with overweight or obesity (OASIS 1): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Aug 26;402(10403):705-719. doi: 10.1016/S0140-6736(23)01185-6. Epub 2023 Jun 26. PMID 37385278